CLINICAL TRIAL: NCT00089622
Title: Transcutaneous Lisuride Therapy of Parkinson's Disease
Brief Title: Lisuride Patch to Treat Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040258; 04-N-0258
Record Dates: First submitted 2004-08-06; First posted 2004-08-09 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-03-31

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Motor Fluctuations; Intravenous Levodopa; Antiparkinsonian Response; Lisuride Patch; Parkinson Disease; PD
MeSH Terms: conditions — Parkinson Disease

INTERVENTIONS:
Drug: Intravenous Levodopa
Drug: Lisuride Transdermal System

SUMMARY:
This study will evaluate the effectiveness of a skin patch formulation of the dopamine agonist Lisuride in controlling parkinsonian symptoms and dyskinesias (involuntary movements) caused by levodopa. Lisuride is currently available in tablet form; this study will test whether a patch formulation that provides continuous stimulation of the dopamine receptors will better control disease symptoms.

Patients between 40 and 80 years old with Parkinson's disease and dyskinesias may be eligible for this 4-month study. Participants undergo the following procedures:

Screening and baseline evaluation: Participants are evaluated with a medical history, physical examination, neurologic evaluation, blood tests, urinalysis, and electrocardiogram. A chest X-ray and MRI or CT scan of the brain are done, if needed. If possible, patients stop taking all antiparkinsonian medications except levodopa (Sinemet) for 1 month (2 months for Selegiline) before the study begins and throughout its duration.

Dose-finding phase: Patients are admitted to the NIH Clinical Center for 2 to 3 days for a levodopa "dose-finding" procedure. For this test, patients stop taking Sinemet and instead have levodopa infused through a vein. During the infusions, the drug dose is increased slowly until parkinsonian symptoms improve or unacceptable side effects occur or the maximum study dose is reached. Symptoms are monitored frequently. (Patients who have had dosing infusions in the last 3 months do not have to undergo this phase of the study.)

Active study phase: Patients are randomly assigned to one of two treatment groups. One group receives a placebo (a patch with no active drug) and a patch that contains Lisuride; the other group receives placebo throughout the entire study. Patients are instructed on how to apply the patches. During the first 2 weeks of this study phase, the number of patches containing active drug is gradually increased until the individual's optimum dose is reached. Patches are changed about every 2 days. During this time, intake of other antiparkinsonian medications is tapered down and patients are evaluated frequently. For the next 3 months, patients wear the patches continuously at the optimum dose. The patches are changed every 2 days or once a week, depending on the individual patient's need. Two levodopa infusion studies are done in the active study phase as they were in the dose-finding phase - at the beginning of the dose escalation phase and again at the end of the dose maintenance phase. In addition, patients are tested for their ability to perform different motor tasks.

Sleep studies: Because oral Lisuride can cause excessive sleepiness, some patients are asked to participate in a sleep study to evaluate sleep patterns during the night and daytime sleepiness. The subject's brain, muscles, and breathing are continuously monitored during sleep. Also, an electroencephalogram (EEG) is done to record brain waves while the subject lies quietly, breathes deeply, watches flashes of light, sleeps, or performs a task.

Safety checks: Patients are monitored closely for safety with a history of side effects, blood tests, and ECG each time a new supply of study drug is dispensed.

Follow-up: 2 weeks after completing the active phase of the study, patients are contacted by phone for a follow-up evaluation.

DETAILED DESCRIPTION:
Introduction: Parkinson's disease (PD) is a progressive degenerative disease of unknown etiology. Treatment is symptomatic and the most successful approach has been to replace the missing dopamine through administration of its precursor levodopa. As the disease progresses, the usefulness of this approach gradually diminishes, and motor complications become a source of significant disability. Although a number of pharmacological strategies have attempted to improve this situation, none has yet proven fully satisfactory. A novel transcutaneous formulation of the dopamine agonist lisuride will be used to test the ability of this approach to reduce levodopa-induced motor response complications.

Objective: The objective of this study is to evaluate the risks and benefits of continuous dopaminomimetic replacement therapy in patients with advanced Parkinson's disease.

Study population: Approximately 22 moderately advanced parkinsonian patients will be enrolled into a randomized, placebo-controlled, double-blind, proof-of-principle study, lasting approximately 16 weeks. Lisuride efficacy will be assessed through the use of validated motor function scales. Safety will be monitored by means of frequent clinical evaluations and laboratory tests.

Anticipated Risks and Benefits: The potential risks associated with this study amount to only a minor increase over minimal risk and are primarily associated with adverse reactions to the medications involved. Lisuride has been approved for use in Europe for more than 20 years and has a wide margin of safety. Patients receiving drug could benefit from improvement of their clinical condition; those on placebo will also receive proper medical care that may lead to a better quality of life.

Outcome Estimate and Potential Meaning for the Field: This study should further the understanding of mechanisms contributing to motor disability in patients with PD and thus lead to the development of improved therapeutic interventions for this disorder and for associated motor response complications.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals who meet all of the following inclusion criteria will be eligible to participate:

Patient has been diagnosed with idiopathic Parkinson's disease.

Patient has relatively advanced disease with levodopa-associated motor response complications, including, peak-dose dyskinesias and wearing-off fluctuations.

Patient can be optimized on oral levodopa, usually with an interdose interval of less than or equal to 3.0 hours.

Patient is willing to adhere to protocol requirements as evidenced by written, informed consent.

Patient is between the ages of 40 and 80 years, inclusive.

EXCLUSION CRITERIA:

Individuals meeting any of the following exclusion criteria immediately before or during the study will not be enrolled or will be immediately excluded from the study, as appropriate:

Patient has a history of any medical condition that can reasonably be expected to subject them to unwarranted risk, such as history of severe cardiac (myocardial infarction within 12 months prior to study, dysrhythmia), severe cerebrovascular, convulsive, significant hepatic (enzyme elevation greater than twice the upper limit of normal), or renal (creatinine exceeding the upper limit of normal) disorder.

Patient is taking a prohibited medication.

Patient is unable to be treated with levodopa/carbidopa alone while a participant in this protocol.

Patient has unilateral or bilateral deep brain stimulating (DBS) devices who are unable or unwilling to turn them off during the period of protocol participation.

Patient has prior bilateral pallidotomy.

Patient has cognitive impairment as indicated by a Minimental status examination (MMSE) score less than 25.

Patient has not been using an adequate contraceptive method for the last 2 months, or (if female) is pregnant or breastfeeding, or not at least one year post-menopausal or unwilling or unable to continue contraceptive use during the study.

Patient has participated in a clinical study with an investigational drug within the last 30 days.

Patient has dermatological problems, such as eczema or hirsutism, that would interfere with transcutaneous therapy.

Patients with known hypersensitivity to lisuride or to skin patch materials.

Patients with slow lisuride metabolism due to CYP450 2D6 deficiency or requiring drugs also metabolized by CYP450 2D6, including Beta-blockers: S-metoprolol, propafenone, antidepressants: amitriptyline, clomipramine, desipramine, imipramine, antipsychotics: haloperidol, risperidone, thioridazine, other drug: codeine, dextromethorphan, flecainide, ondansetron, and tramadol.

CONCOMITANT MEDICATION EXCLUSION:

The following medications are prohibited for at least one month prior to randomization (except as noted below) and during the course of study:

Dopamine agonists of any kind (for 1 week, Cabergoline for 8 weeks).

Any investigational drug not specifically permitted in the protocol.

MAO inhibitors, such as selegiline (for 2 months).

Anticholinergics.

Drugs not used primarily to treat Parkinson's disease but which may modify parkinsonian symptoms, including neuroleptics, metoclopramide and alpha or beta adrenergic receptor antagonists.

Drugs considered to ameliorate dyskinesias including NMDA antagonists (such as amantadine, budipine, memantine, remacemide and dextromethorphan), alpha or beta adrenergic receptor antagonists, anxiolytics (such as buspirone) with the exception of antidepressants from the SSRI group such as fluoxetine, antipsychotics (such as clozapine, quetiapine and olanzapine), cannabinoid receptor antagonists, and adenosine A2a antagonists, or to exacerbate dyskinesias (such as sodium valproate and CNS stimulants).

Drugs known to have 5HT receptor subtype affinity (such as ritanserin, sumatriptan).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-08-04; Study Completion 2007-03-31

PRIMARY OUTCOMES:
Change in parkinsonian severity variance.

SECONDARY OUTCOMES:
Change in dyskinesia severity.
Change in antiparkinsonian efficacy half-time for levodopa.
Change in parkinsonian severity.
Change in optimal oral levodopa requirement.
Change in patient diary rating.
Change in daytime somnolence.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Grace AA, Bunney BS. The control of firing pattern in nigral dopamine neurons: single spike firing. J Neurosci. 1984 Nov;4(11):2866-76. doi: 10.1523/JNEUROSCI.04-11-02866.1984. PMID 6150070